CLINICAL TRIAL: NCT05185362
Title: Retrospective Study on Pecan Nut Allergy Epidemiology
Brief Title: Epidemiology of Pecan Nut Allergy
Acronym: PEC-ALL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0726
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Allergic Reaction
Keywords: Sensitization to pecan nut (specific IgE and/or skin prick tests); Challenge proven pecan allergy; Allergic Comorbidities; Oral food challenge; Anaphylaxis
MeSH Terms: conditions — Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IgE-mediated food allergy can manifest with reactions ranging from hives to anaphylactic shock. The diagnosis is based on the confirmation of sensitization to the food allergen by skin tests (prick) and the determination of specific IgE directed against the food source and molecular allergens. The gold standard remains the oral provocation test, which is performed in a hospital environment. Once the diagnosis is made, an elimination diet is still considered as the cornerstone of treatment for most food allergies.

While some allergies, such as cow's milk or egg, tend to resolve spontaneously, others, such as allergy to pecan nuts, show a tendency to be persistent. In addition, pecan allergy is often characterized by potentially serious clinical reactions, compared to other foods, which can even be life threatening. In our clinical practice, the investigators found that patients with allergies to pecan nuts often present with severe hypersensitivity reactions when challenged orally to this food. Beyond this information, there are few studies regarding pecans. The investigators decided to retrospectively evaluate the results of oral food challenge and of the allergy work-up in our patients sensitized and allergic to pecan nuts, to better understand the current epidemiology of such food allergy.

ELIGIBILITY:
Inclusion criteria:

* Patients assessed for pecan allergy, through oral food challenge, from January 2000 to december 2021, at the University Hospital of Montpellier
* Patients with a positive skin prick test and/or positive specific IgE to pecan nut

Exclusion criteria:

* Patients not affiliated to French Social Security
* Patients not capable of understanding French
* Patients sensitized to pecan nut, who did not perform an oral food challenge to this food allergen

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting in the Allergy Unit of the Arnaud de Villeneuve Hospital, sensitized to pecan nut, and having undergone an oral food challenge to this food allergen
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of challenge-proven pecan allergy | day 1
  Prevalence of challenge-proven pecan allergy in sensitized patients

SECONDARY OUTCOMES:
Epidemiological characteristics of pecan allergic patient | day 1
  Epidemiological characteristics of pecan allergic patient(cypress pollen-induced allergic rhinitis or food allergy to peach)
cut-off of specific IgE | day 1
  cut-off of specific IgE and of results of prick test to predict pecan allergy in sensitized and allergic patients

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC